CLINICAL TRIAL: NCT00760474
Title: A Double-Blind, Placebo-Controlled Cross-Over Study In Fibromyalgia Subjects To Examine Effects Of Pregabalin On Brain Response To Mechanical Pain As Assessed By Functional Magnetic Resonance Imaging, Proton Magnetic Resonance Spectroscopy And Subjective Ratings
Brief Title: An fMRI Study Of Brain Response In Patients With Fibromyalgia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: A0081211
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Results first posted 2012-04-04 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2018-11

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; fMRI; pain; pregabalin; Lyrica; imaging
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin, then placebo (Experimental)
  Interventions: Drug: Pregabalin, then placebo
- Placebo, then pregabalin (Experimental)
  Interventions: Drug: Placebo, then pregabalin

INTERVENTIONS:
Drug: Pregabalin, then placebo — Placebo and pregabalin will be given orally twice daily in capsules at different times during the course of the study. The highest dose of pregabalin to be used in the study is 450 mg/day.
  Arms: Pregabalin, then placebo
Drug: Placebo, then pregabalin — Placebo and pregabalin will be given orally twice daily in capsules at different times during the course of the study. The highest dose of pregabalin to be used in the study is 450 mg/day.
  Arms: Placebo, then pregabalin

SUMMARY:
The purpose of this study is to explore how pregabalin works in patients with fibromyalgia by evaluating brain imaging signals. To find out whether fMRI (functional magnetic resonance imaging) is an efficient way to show whether new pain medications are effective in treating fibromyalgia.

DETAILED DESCRIPTION:
Methodology study

ELIGIBILITY:
Inclusion Criteria:

* Women must have pain due to fibromyalgia
* Fibromyalgia must have been diagnosed at least 6 months prior to be eligible for this study

Exclusion Criteria:

* Patients with severe depression or other serious illness, who are left-handed, or who are pregnant or nursing are not eligible for this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Ichesco E, Peltier SJ, Mawla I, Harper DE, Pauer L, Harte SE, Clauw DJ, Harris RE. Prediction of Differential Pharmacologic Response in Chronic Pain Using Functional Neuroimaging Biomarkers and a Support Vector Machine Algorithm: An Exploratory Study. Arthritis Rheumatol. 2021 Nov;73(11):2127-2137. doi: 10.1002/art.41781. Epub 2021 Sep 22. PMID 33982890
- [Derived] Puiu T, Kairys AE, Pauer L, Schmidt-Wilcke T, Ichesco E, Hampson JP, Napadow V, Clauw DJ, Harris RE. Association of Alterations in Gray Matter Volume With Reduced Evoked-Pain Connectivity Following Short-Term Administration of Pregabalin in Patients With Fibromyalgia. Arthritis Rheumatol. 2016 Jun;68(6):1511-21. doi: 10.1002/art.39600. PMID 26816332
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081211&StudyName=An%20fMRI%20Study%20Of%20Brain%20Response%20In%20Patients%20With%20Fibromyalgia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who met entrance criteria received placebo for 1 week (Day 1 to 8) then were randomized in a 1:1 ratio to blinded treatment sequence.
Groups:
- Pregabalin First, Then Placebo: Pregabalin 75 milligrams (mg) by mouth (PO) twice daily (BID) Period 1/Day 9 to 11; 150 mg BID Day 12 to 16; 200 mg BID Day 17 to 19; 225 mg BID Day 20 to 22 followed by taper Day 23 to 29 and an 8-day placebo washout period. Then, placebo matching study treatment in a similar pattern was administered beginning Period 2/Day 38.
- Placebo First, Then Pregabalin: Placebo matching study treatment was administered beginning Period 1/Day9. Then, Pregabalin 75 mg BID Period 2/Day 38 to 40; 150 mg BID Day 41 to 45; 200 mg BID Day 46 to 48; 225 mg BID Day 49 to 51 followed by placebo taper Day 52 to 58.
Period: Period 1 (P1)
Arm/Group | Pregabalin First, Then Placebo | Placebo First, Then Pregabalin
Started | 13 | 14
Treated | 13 (1 participant discontinued in P1; re-entered with new identification number and completed P1, P2.) | 14 (1 participant discontinued in P1; re-entered with new identification number and completed P1, P2.)
Overall Number of Unique Participants | 12 | 13
Completed | 12 | 13
Not Completed | 1 | 1
Not completed — Discontinued then re-entered | 1 | 1
Period: Placebo Washout Period
Arm/Group | Pregabalin First, Then Placebo | Placebo First, Then Pregabalin
Started | 12 | 13
Completed | 12 | 12
Not Completed | 0 | 1
Not completed — Other | 0 | 1
Period: Period 2 (P2)
Arm/Group | Pregabalin First, Then Placebo | Placebo First, Then Pregabalin
Started | 12 | 12
Completed | 11 | 11
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Participants who met entrance criteria received placebo for 1 week (Day 1 to 8) then were randomized in a 1:1 ratio to blinded treatment sequence to receive either:
  Pregabalin, then placebo: Pregabalin 75 mg PO BID Period 1/Day 9 to 11; 150 mg BID Day 12 to 16; 200 mg BID Day 17 to 19; 225 mg BID Day 20 to 22 followed by taper Day 23 to 29 and an 8-day placebo washout period. Then, placebo matching study treatment in a similar pattern was administered beginning Period 2/Day 38 and included dose escalation through Day 51 followed by placebo taper Day 52 to 58.
  Or placebo, then Pregabalin: Placebo matching study treatment was administered in a similar fashion to Pregabalin treatment beginning Period 1/Day 9 and included dose escalation, taper and an 8-day placebo washout period. Then, Pregabalin 75 mg BID Period 2/Day 38 to 40; 150 mg BID Day 41 to 45; 200 mg BID Day 46 to 48; 225 mg BID Day 49 to 51 followed by placebo taper Day 52 to 58.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (12.0)
Sex/Gender, Customized [Number; unit: participants] — Female
  participants | 25

OUTCOME MEASURES:

1. Primary Outcome: Glutamine/Creatine (Gln/Cr) and Glutamate/Creatine (Glu/Cr) Ratios Measured by Proton Magnetic Resonance Spectroscopy (1H-MRS)
Description: Single voxel spectra obtained from the anterior and posterior right insula at rest to compare ratios for Gln/Cr, Glu/Cr, and combined Glutamate + Glutamine (Glx/Cr) for pregabalin and placebo. Gln, Glu, Glx calculated as ratios to the internal standard creatine.
Time Frame: Baseline (Day 8, Day 37), Post-dose (Period 1/Day 22, Period 2/Day 51)
Population: Full Analysis Set (FAS) all participants who received a minimum fixed dose of 300 mg/day of study treatment. N=number of participants with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Pregabalin: Pregabalin administered in Period 1 (75 mg BID Period 1/Day 9 to 11; then 150 mg BID Period 1/Day 12 to 16; then 200 mg BID Period 1/Day 17 to 19; then 225 mg BID Period 1/Day 20 to 22) or administered in Period 2 (75 mg BID Period 2/Day 38 to 40; then 150 mg BID Period 2/Day 41 to 45; then 200 mg BID Period 2/Day 46 to 48; then 225 mg BID Period 2/Day 49 to 51); then taper Period 2/Day 52 to 58.
- Placebo: Placebo to match study treatment administered in Period 1 or Placebo to match study treatment administered in Period 2.
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 17 | 17
ratio
  Glu/Cr ratio posterior insula - pre-dose | 1.1751 (0.119537) | 1.13253 (0.123897)
  Glu/Cr ratio posterior insula - post-dose | 1.1046 (0.14180) | 1.17129 (0.151535)
  Gln/Cr ratio posterior insula - pre-dose | 0.5311 (0.117359) | 0.52635 (0.143649)
  Gln/Cr ratio posterior insula - post-dose | 0.4857 (0.14534) | 0.51553 (0.147882)
  Glx/Cr ratio posterior insula - pre-dose | 1.70624 (0.177312) | 1.65894 (0.215505)
  Glx/Cr ratio posterior insula - post-dose | 1.5903 (0.19461) | 1.68747 (0.227398)
  Glu/Cr ratio anterior insula - pre-dose | 1.22731 (0.154333) | 1.23788 (0.183282)
  Glu/Cr ratio anterior insula - post-dose | 1.2393 (0.22290) | 1.18524 (0.164847)
  Gln/Cr ratio anterior insula - pre-dose | 0.53144 (0.115606) | 0.47882 (0.143684)
  Gln/Cr ratio anterior insula - post-dose | 0.5290 (0.19367) | 0.47541 (0.100247)
  Glx/Cr ratio anterior insula - pre-dose | 1.75888 (0.164256) | 1.71671 (0.203157)
  Glx/Cr ratio anterior insula - post-dose | 1.7684 (0.30019) | 1.66124 (0.166421)
Statistical Analysis 1: Comparison: Pregabalin; Glu/Cr posterior insula; Test type: Superiority or Other; p = 0.083, t-test, 2 sided — Significance was set at p <0.05; Mean Difference (Final Values) = -0.070, Standard Deviation 0.157 — Mean difference between the pre-dose (baseline) and post-dose values calculated as post-dose minus pre-dose (post minus pre)
Statistical Analysis 2: Comparison: Placebo; Glu/Cr posterior insula; Test type: Superiority or Other; p = 0.436, t-test, 2 sided — Significance was set at p <0.05
Statistical Analysis 3: Comparison: Pregabalin; Gln/Cr posterior insula; Test type: Superiority or Other; p = 0.306, t-test, 2 sided; Significance was set at p <0.05
Statistical Analysis 4: Comparison: Placebo; Gln/Cr posterior insula; Test type: Superiority or Other; p = 0.809, t-test, 2 sided; Significance was set at p <0.05
Statistical Analysis 5: Comparison: Pregabalin; Glx/Cr posterior insula; Test type: Superiority or Other; p = 0.016, t-test, 2 sided; Significance was set at p <0.05; Mean Difference (Final Values) = -0.116, Standard Deviation 0.177 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Placebo; Glx/Cr posterior insula; Test type: Superiority or Other; p = 0.708, t-test, 2 sided — Significance was set at p <0.05; Mean Difference (Final Values) = 0.029, Standard Deviation 0.308 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Pregabalin; Glu/Cr anterior insula; Test type: Superiority or Other; p = 0.809, t-test, 2 sided — Significance was set at p <0.050
Statistical Analysis 8: Comparison: Placebo; Glu/Cr anterior insula; Test type: Superiority or Other; p = 0.154, t-test, 2 sided — Significance was set at p <0.05
Statistical Analysis 9: Comparison: Pregabalin; Gln/Cr anterior insula; Test type: Superiority or Other; p = 0.960, t-test, 2 sided; Significance was set at p <0.05
Statistical Analysis 10: Comparison: Placebo; Gln/Cr anterior insula; Test type: Superiority or Other; p = 0.937, t-test, 2 sided; Significance was set at p <0.05
Statistical Analysis 11: Comparison: Pregabalin; Glx/Cr anterior insula; Test type: Superiority or Other; p = 0.897, t-test, 2 sided — Significance was set at p <0.05
Statistical Analysis 12: Comparison: Placebo; Glx/Cr anterior insula; Test type: Superiority or Other; p = 0.309, t-test, 2 sided — Significance was set at p <0.05

2. Primary Outcome: Voxel-wise Blood Oxygen Level Dependent (BOLD) Using Functional Magnetic Resonance Imaging (fMRI) of Brain Activation Signals in Response to Blunt Pressure Pain: Percent Change in BOLD Activations Including Outliers
Description: BOLD fMRI imaging modality to assess brain activation signals across the whole brain in defined Region of Interest (ROI) brain regions in response to blunt pressure pain; acquired during resting state (no evoked pain) and during evoked pain (thumb pressure device with non-painful pressure, 2 kilograms [kg] pressure/equal stimulus conditions, and high pain pressure/up to 10 kg). Estimated as magnitude (percent change) of the betas representing brain signal activation associated with pressure induced pain. Any observation with a studentized residual >3 or <-3 was considered an outlier.
Time Frame: Baseline (Day 8, Day 37), Post-dose (Period 1/Day 22, Period 2/Day 51)
Population: FAS. Change from baseline for Period 1 and Period 2 summarized as Least Squares Mean (LS Mean). Abbreviation: Dorso Lateral Prefrontal Cortex (DLPFC).
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 16 | 16
percent change
  Anterior Cingulate | 0.008 (0.0454) | -0.024 (0.0454)
  Brodman Area (BA) 22 | -0.050 (0.0709) | 0.029 (0.0709)
  BA40 | -0.047 (0.0436) | 0.026 (0.0436)
  Left (L)_Anterior Insula (anIns) | 0.073 (0.0378) | 0.044 (0.0378)
  L_Amygdala | -0.040 (0.0502) | 0.041 (0.0502)
  L_Cerebellum | -0.056 (0.0317) | 0.021 (0.0317)
  L_DLPFC | -0.002 (0.0255) | 0.023 (0.0255)
  L_Mid Insula | -0.011 (0.0672) | 0.100 (0.0672)
  L_Mid Temporal Pole | -0.024 (0.0307) | -0.044 (0.0307)
  L_Orbito Front | 0.033 (0.1000) | -0.136 (0.1000)
  Periaqueductal gray (PAG) | 0.014 (0.0351) | 0.016 (0.0351)
  Posterior Insula (pIns) | 0.001 (0.0294) | 0.002 (0.0294)
  L_Posterior Cingulate | -0.132 (0.0414) | -0.083 (0.0414)
  L_Precuneus | -0.057 (0.0281) | -0.084 (0.0281)
  L_Putamen | 0.081 (0.0347) | 0.037 (0.0347)
  L_Secondary Somatosensory Area (S2) | -0.016 (0.0746) | 0.111 (0.0746)
  Right (R)_DLPFC | -0.004 (0.0467) | 0.101 (0.0467)
  R_Anterior Insula | 0.080 (0.0378) | 0.002 (0.0378)
  R_Amygdala | -0.077 (0.0572) | 0.076 (0.0572)
  R_BA23_base | 0.005 (0.0267) | -0.017 (0.0267)
  R_Inferior Parietal Lobule (IPL)_base | -0.042 (0.0301) | -0.015 (0.0301)
  R_Insula_base | -0.010 (0.0595) | 0.034 (0.0595)
  R_Mid Insula | 0.015 (0.0423) | 0.028 (0.0423)
  R_Mid Front_DLPFC | -0.011 (0.0432) | 0.083 (0.0432)
  R_Mid Temporal Pole | -0.048 (0.0250) | -0.036 (0.0250)
  R_Orbito Front | -0.046 (0.0709) | -0.056 (0.0709)
  L_PAG | 0.034 (0.0349) | 0.011 (0.0349)
  R_Posterior Insula | 0.063 (0.0345) | -0.024 (0.0345)
  Posterior Insula | 0.050 (0.0434) | -0.002 (0.0434)
  R_Posterior Cingulate | -0.175 (0.0476) | -0.093 (0.0476)
  R_Precuneus | -0.070 (0.0332) | -0.070 (0.0332)
  R_Precuneus_base | -0.040 (0.0273) | -0.038 (0.0273)
  Superior Temporal | -0.039 (0.0645) | 0.026 (0.0645)
  R_Premotor | -0.022 (0.0415) | -0.022 (0.0415)
  R_Putamen | 0.088 (0.0395) | 0.032 (0.0395)
  R_Primary Somatosensory Area (S1) | -0.048 (0.0419) | 0.037 (0.0419)
  R_Thalamus | 0.010 (0.0245) | 0.018 (0.0245)
  Precuneus | -0.066 (0.0301) | -0.078 (0.0301)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Anterior Cingulate; Test type: Superiority or Other; p = 0.6347, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = 0.032, 95% CI 2-sided [-0.1081 to 0.1714]
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; BA22; Test type: Superiority or Other; p = 0.5181, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.079, 95% CI 2-sided [-0.3356 to 0.1771]
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; BA40; Test type: Superiority or Other; p = 0.2987, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.072, 95% CI 2-sided [-0.2161 to 0.0714]
Statistical Analysis 4: Comparison: Pregabalin vs Placebo; L_anIns; Test type: Superiority or Other; p = 0.5151, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = 0.029, 95% CI 2-sided [-0.0640 to 0.1219]
Statistical Analysis 5: Comparison: Pregabalin vs Placebo; L_Amygdala; Test type: Superiority or Other; p = 0.2369, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.081, 95% CI 2-sided [-0.2228 to 0.0599]
Statistical Analysis 6: Comparison: Pregabalin vs Placebo; L_Cerebellum; Test type: Superiority or Other; p = 0.0758, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.077, 95% CI 2-sided [-0.1642 to 0.0092]
Statistical Analysis 7: Comparison: Pregabalin vs Placebo; L_DLPFC; Test type: Superiority or Other; p = 0.4609, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.025, 95% CI 2-sided [-0.0947 to 0.0452]
Statistical Analysis 8: Comparison: Pregabalin vs Placebo; L_Mid Insula; Test type: Superiority or Other; p = 0.3813, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.111, 95% CI 2-sided [-0.3745 to 0.1524]
Statistical Analysis 9: Comparison: Pregabalin vs Placebo; L_Mid Temporal Pole; Test type: Superiority or Other; p = 0.7200, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = 0.020, 95% CI 2-sided [-0.0964 to 0.1361]
Statistical Analysis 10: Comparison: Pregabalin vs Placebo; L_Orbito Front; Test type: Superiority or Other; p = 0.2099, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = 0.168, 95% CI 2-sided [-0.1065 to 0.4434]
Statistical Analysis 11: Comparison: Pregabalin vs Placebo; PAG; Test type: Superiority or Other; p = 0.9551, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.003, 95% CI 2-sided [-0.1047 to 0.0992]
Statistical Analysis 12: Comparison: Pregabalin vs Placebo; Posterior Insula; Test type: Superiority or Other; p = 0.9940, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.000, 95% CI 2-sided [-0.0855 to 0.0848]
Statistical Analysis 13: Comparison: Pregabalin vs Placebo; L_Posterior Cingulate; Test type: Superiority or Other; p = 0.4291, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.049, 95% CI 2-sided [-0.1792 to 0.0806]
Statistical Analysis 14: Comparison: Pregabalin vs Placebo; L_Precuneus; Test type: Superiority or Other; p = 0.4670, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = 0.027, 95% CI 2-sided [-0.0496 to 0.1028]
Statistical Analysis 15: Comparison: Pregabalin vs Placebo; L_Putamen; Test type: Superiority or Other; p = 0.4443, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = 0.044, 95% CI 2-sided [-0.0752 to 0.1624]
Statistical Analysis 16: Comparison: Pregabalin vs Placebo; L_S2; Test type: Superiority or Other; p = 0.2823, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.127, 95% CI 2-sided [-0.3704 to 0.1165]
Statistical Analysis 17: Comparison: Pregabalin vs Placebo; R_DLPFC; Test type: Superiority or Other; p = 0.1369, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.105, 95% CI 2-sided [-0.2481 to 0.0378]
Statistical Analysis 18: Comparison: Pregabalin vs Placebo; R_anIns; Test type: Superiority or Other; p = 0.2376, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = 0.078, 95% CI 2-sided [-0.0573 to 0.2127]
Statistical Analysis 19: Comparison: Pregabalin vs Placebo; R_Amygdala; Test type: Superiority or Other; p = 0.0968, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.153, 95% CI 2-sided [-0.3365 to 0.0313]
Statistical Analysis 20: Comparison: Pregabalin vs Placebo; R_BA23_base; Test type: Superiority or Other; p = 0.5720, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = 0.023, 95% CI 2-sided [-0.0610 to 0.1062]
Statistical Analysis 21: Comparison: Pregabalin vs Placebo; R_IPL_base; Test type: Superiority or Other; p = 0.5822, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.027, 95% CI 2-sided [-0.1303 to 0.0761]
Statistical Analysis 22: Comparison: Pregabalin vs Placebo; R_Insula_base; Test type: Superiority or Other; p = 0.6851, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.044, 95% CI 2-sided [-0.2697 to 0.1824]
Statistical Analysis 23: Comparison: Pregabalin vs Placebo; R_Mid Insula; Test type: Superiority or Other; p = 0.8656, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.013, 95% CI 2-sided [-0.1699 to 0.1446]
Statistical Analysis 24: Comparison: Pregabalin vs Placebo; R_Mid Front_DLPFC; Test type: Superiority or Other; p = 0.1562, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.094, 95% CI 2-sided [-0.2296 to 0.0407]
Statistical Analysis 25: Comparison: Pregabalin vs Placebo; R_Mid Temporal Pole; Test type: Superiority or Other; p = 0.7752, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.012, 95% CI 2-sided [-0.0991 to 0.0754]
Statistical Analysis 26: Comparison: Pregabalin vs Placebo; R_Orbito Front; Test type: Superiority or Other; p = 0.9182, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = 0.010, 95% CI 2-sided [-0.1912 to 0.2109]
Statistical Analysis 27: Comparison: Pregabalin vs Placebo; L_PAG; Test type: Superiority or Other; p = 0.6544, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = 0.022, 95% CI 2-sided [-0.0829 to 0.1278]
Statistical Analysis 28: Comparison: Pregabalin vs Placebo; R_pIns; Test type: Superiority or Other; p = 0.0813, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = 0.087, 95% CI 2-sided [-0.0123 to 0.1863]
Statistical Analysis 29: Comparison: Pregabalin vs Placebo; R_pIns; Test type: Superiority or Other; p = 0.4605, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = 0.052, 95% CI 2-sided [-0.0956 to 0.2004]
Statistical Analysis 30: Comparison: Pregabalin vs Placebo; R_Posterior Cingulate; Test type: Superiority or Other; p = 0.3136, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.081, 95% CI 2-sided [-0.2484 to 0.0856]
Statistical Analysis 31: Comparison: Pregabalin vs Placebo; R_Precuneus; Test type: Superiority or Other; p = 0.9929, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = 0.000, 95% CI 2-sided [-0.0885 to 0.0893]
Statistical Analysis 32: Comparison: Pregabalin vs Placebo; R_Precuneus_base; Test type: Superiority or Other; p = 0.9490, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.002, 95% CI 2-sided [-0.0815 to 0.0767]
Statistical Analysis 33: Comparison: Pregabalin vs Placebo; Superior Temporal; Test type: Superiority or Other; p = 0.5668, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.065, 95% CI 2-sided [-0.3019 to 0.1722]
Statistical Analysis 34: Comparison: Pregabalin vs Placebo; R_Premotor; Test type: Superiority or Other; p = 0.9958, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.000, 95% CI 2-sided [-0.1398 to 0.1391]
Statistical Analysis 35: Comparison: Pregabalin vs Placebo; R_Putamen; Test type: Superiority or Other; p = 0.3379, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = 0.057, 95% CI 2-sided [-0.0659 to 0.1795]
Statistical Analysis 36: Comparison: Pregabalin vs Placebo; R_S1; Test type: Superiority or Other; p = 0.2186, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.085, 95% CI 2-sided [-0.2262 to 0.0565]
Statistical Analysis 37: Comparison: Pregabalin vs Placebo; R_Thalamus; Test type: Superiority or Other; p = 0.8191, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = -0.008, 95% CI 2-sided [-0.0843 to 0.0678]
Statistical Analysis 38: Comparison: Pregabalin vs Placebo; Precuneus; Test type: Superiority or Other; p = 0.7647, Mixed Models Analysis — Significance was set at p <0.05; Mixed-effect repeated measure model included participant as a random effect; treatment, visit as fixed effects; Least Squares (LS) Mean difference = 0.012, 95% CI 2-sided [-0.0698 to 0.0930]

3. Secondary Outcome: Voxel-wise Blood Oxygen Level Dependent (BOLD) Using Functional Magnetic Resonance Imaging (fMRI) of Brain Activation Signals in Response to a Control Visual (Checkerboard) Stimuli
Description: BOLD fMRI imaging modality to assess brain activation signals across the whole brain in defined ROI brain regions in response to checkerboard visual stimuli (flashing at 8 hertz [Hz]). Reported as percent change between the pre-dose (baseline) and post-dose values.
Time Frame: Baseline (Day 8, Day 37), Post-dose (Period 1/Day 22, Period 2/Day 51)
Population: FAS.
Measure: Mean (Standard Deviation); unit: percent change in BOLD signal
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 17 | 17
percent change in BOLD signal
  Right (R) anterior mid insula cortex | 0.32 (0.19) | -0.05 (0.25)
  Left (L) mid insula cortex | 0.23 (0.20) | 0.00 (0.21)
  R inferior parietal lobule, Brodman area 40 | 0.27 (0.21) | 0.05 (0.23)
  L inferior parietal lobule, Brodman area 40 | 0.28 (0.27) | 0.02 (0.25)
  Right primary somatosensory cortex | 0.14 (0.14) | -0.01 (0.22)
  Left primary somatosensory cortex | 0.21 (0.18) | 0.06 (0.25)
  Left supplementary motor area | 0.02 (0.32) | 0.30 (0.34)

4. Secondary Outcome: Resting State Brain Activity (Connectivity Analysis) Assessed by Temporal Correlations in Low Frequency fMRI BOLD Signals Across Pain Processing Regions
Description: Resting state brain activity assessed for correlation of brain seed region (pIns, anIns) to ROI connectivity at baseline (pre-dose) and post-dose (pre minus post) measured using z-score (mean of 0, standard deviation [SD] of 1); range approximately -3 to +3. Positive (+) z-scores reflect greater connectivity (+correlation between seed region and ROI). Negative (-) z-scores reflect -connectivity (anti-correlation between seed region and ROI). ROIs include PCC and IPL from within the default mode network (DMN). DMN is a constellation of regions in which connectivity is augmented in fibromyalgia.
Time Frame: Baseline (Day 8, Day 37), Post-dose (Period 1/Day 22, Period 2/Day 51)
Population: Participants in FAS with quality resting state data (data able to be corrected for motion [head and cardiorespiratory artifacts]).
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 14 | 14
z-score
  pIns_Posterior cingulate (PCC) pre-dose | 1.1647 (1.71738) | 1.5405 (1.70926)
  pIns_PCC post-dose | 2.1504 (1.87564) | 1.2409 (2.29890)
  pIns_primary motor region (M1) pre-dose | 3.1486 (3.14585) | 1.3267 (1.94564)
  pIns_M1 post-dose | 3.2605 (2.80878) | 1.3771 (2.01620)
  pIns_cerebellum pre-dose | 0.3984 (1.73000) | 1.4439 (1.46341)
  pIns_cerebellum post-dose | 0.0213 (2.24014) | 1.0704 (2.66882)
  pIns_Left (L) IPL 3a pre-dose | 0.2025 (1.92233) | -0.9296 (1.50499)
  pIns_L IPL 3a post-dose | -0.3792 (2.18759) | -1.2977 (1.37551)
  pIns_L IPL 3b pre-dose | 0.6552 (1.82208) | 1.7390 (2.00764)
  pIns_L IPL 3b post-dose | 1.5614 (1.58417) | 0.9930 (2.50930)
  pIns_Right (R) IPL 3b pre-dose | 0.8310 (2.01819) | 0.7420 (1.57551)
  pIns_R IPL 3b post-dose | 0.9766 (2.52679) | 0.9081 (2.18440)
  pIns_cuneus pre-dose | 2.1363 (1.97131) | 1.8543 (1.85494)
  pIns_cuneus post-dose | 3.0410 (1.84499) | 2.3324 (1.84622)
  anIns_L IPL pre-dose | 2.1404 (2.21726) | 1.9982 (2.40790)
  anIns_L IPL post-dose | 2.6493 (2.04040) | 2.6797 (2.50765)
  anIns_R IPL pre-dose | 2.6956 (2.61359) | 1.7848 (2.27345)
  anIns_R IPL post-dose | 1.2863 (1.31165) | 2.6194 (2.37251)
  anIns_S2 pre-dose | 1.6592 (1.69160) | 1.6799 (1.64784)
  anIns_S2 post-dose | 3.1466 (2.13680) | 2.4225 (2.68238)
  anIns_cuneus pre-dose | 2.5103 (2.48669) | 1.7550 (1.65232)
  anIns_cuneus post-dose | 1.8042 (2.08443) | 1.1899 (1.67701)

5. Secondary Outcome: Gracely Box Scales for Pain Intensity (GBSint) Including Outliers
Description: Minimum and maximum pain intensity acquired during resting state (no evoked pain) and during evoked pain (thumb pressure device with non-painful pressure, 2 kg pressure/equal stimulus conditions, and high pain pressure/up to 10 kg) measured during fMRI and scored from 0 (no pain sensation) to 20 (extremely intense). Baseline and Post-dose data for Period 1 and Period 2 summarized as Least Squares Mean (LS Mean). Any observation with a studentized residual >3 or <-3 was considered an outlier.
Time Frame: Baseline (Day 8, Day 37), Post-dose (Period 1/Day 22, Period 2/Day 51)
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 22 | 22
scores on a scale
  Minimum pain intensity | 4.1184 (0.6535) | 3.4725 (0.6535)
  Maximum pain intensity | 14.5701 (0.6953) | 15.6117 (0.6953)

6. Secondary Outcome: Gracely Box Scales for Pain Unpleasantness (GBSunp) Including Outliers
Description: Minimum and maximum pain unpleasantness acquired during resting state (no evoked pain) and during evoked pain (thumb pressure device with non-painful pressure, 2 kg pressure/equal stimulus conditions, and high pain pressure/up to 10 kg) measured during fMRI and scored from 0 (neutral) to 20 (very intolerable). Baseline and Post-dose data for Period 1 and Period 2 summarized as LS Mean. Any observation with a studentized residual >3 or <-3 was considered an outlier.
Time Frame: Baseline/Pre-dose (Day 8, Day 37), Post-dose (Period 1/Day 22, Period 2/Day 51)
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 22 | 22
scores on a scale
  Minimum pain unpleasantness | 3.3924 (0.5803) | 3.4258 (0.5803)
  Maximum pain unpleasantness | 10.1576 (0.8294) | 11.2742 (0.8294)

7. Secondary Outcome: Daily Pain Diary Numeric Rating Scale (NRS) Item From the Modified Brief Pain Inventory (mBPI) for Assessment of Clinical Pain: 7 Day Average Pain Score Including Outliers
Description: The daily pain diary consisted of the mBPI item regarding participant-rated average of pain over the past 24 hours. Scored on an 11-point numeric scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine). The 7 day average pain score was defined as the mean daily pain NRS value for the last 7 days prior to fMRI scanning visit. Baseline and Post-dose data for Period 1 and Period 2 summarized as LS Mean. Any observation with a studentized residual >3 or <-3 was considered an outlier.
Time Frame: Baseline (Day 8, Day 37), Post-dose (Period 1/Day 22, Period 2/Day 51)
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 22 | 22
scores on a scale | 4.1014 (0.4104) | 4.7038 (0.4104)

8. Secondary Outcome: Daily Pain Diary Numeric Rating Scale (NRS) Item From the Modified Brief Pain Inventory (mBPI) for Assessment of Clinical Pain: 3 Day Average Pain Score Including Outliers
Description: The daily pain diary consisted of the mBPI item regarding participant-rated average of pain over the past 24 hours. Scored on an 11-point numeric scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine). The 3 day average pain score was defined as the mean daily pain NRS value for the last 3 days prior to fMRI scanning visit. Baseline and Post-dose data for Period 1 and Period 2 summarized as LS Mean. Any observation with a studentized residual >3 or <-3 was considered an outlier.
Time Frame: Baseline (Day 8, Day 37), Post-dose (Period 1/Day 22, Period 2/Day 51)
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 22 | 22
scores on a scale | 4.3467 (0.4436) | 4.7745 (0.4436)

9. Secondary Outcome: Daily Pain Diary Numeric Rating Scale (NRS) Item From the Modified Brief Pain Inventory (mBPI) for Assessment of Clinical Pain: Individual Daily Pain Score Including Outliers
Description: The daily pain diary consisted of the mBPI item regarding participant-rated average of pain over the past 24 hours. Scored on an 11-point numeric scale ranging from 0 (no pain) to 10 (pain as bad as you can imagine). The individual daily pain score was defined as the final score recorded in the last pain diary of the treatment period 24 hours prior to fMRI scanning visit. Baseline and Post-dose data for Period 1 and Period 2 summarized as LS Mean. Any observation with a studentized residual >3 or <-3 was considered an outlier.
Time Frame: Baseline (Day 8, Day 37), Post-dose (Period 1/Day 22, Period 2/Day 51)
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 22 | 22
scores on a scale | 4.3110 (0.4787) | 5.0527 (0.4787)

10. Secondary Outcome: Short-Form McGill Pain Questionnaire (SF-MPQ): Affective Total Score Including Outliers
Description: SF-MPQ was completed to assess pain over the past week and to assess present pain and consists of 15 pain descriptors: sensory dimension of pain experience (sum of items 1 to 11) and affective dimension (sum of items 12 to 15). Each descriptor was ranked by participant on a 4-point intensity scale (0=none to 3=severe) and totaled in each subclass (sensory range 0 to 33; affective range 0 to 12); higher scores indicated higher pain/impact. Baseline and Post-dose data for Period 1 and Period 2 summarized as LS Mean. Any observation with a studentized residual >3 or <-3 was considered an outlier.
Time Frame: Baseline (Day 8, Day 37), Post-dose (Period 1/Day 22, Period 2/Day 51)
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 22 | 22
scores on a scale | 1.4100 (0.3095) | 1.8173 (0.3095)

11. Secondary Outcome: Short-Form McGill Pain Questionnaire (SF-MPQ): Sensory Total Score Including Outliers
Description: as for outcome 10
Time Frame: Baseline (Day 8, Day 37), Post-dose (Period 1/Day 22, Period 2/Day 51)
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 22 | 22
scores on a scale | 8.6641 (1.0759) | 9.4722 (1.0759)

12. Other Pre Specified Outcome: Hospital Anxiety and Depression Scale (HADS): Anxiety Total Score Including Outliers
Description: A participant rated questionnaire with 2 subscales. HADS-A assessed state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D assessed state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicated greater severity of anxiety and depression symptoms. Any observation with a studentized residual >3 or <-3 was considered an outlier.
Time Frame: Baseline (Day 8, Day 37), Post-dose (Period 1/Day 22, Period 2/Day 51)
Population: FAS. Baseline and Post-dose data for Period 1 and Period 2 summarized as LS Mean.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 22 | 22
scores on a scale | 4.3896 (0.6132) | 5.1558 (0.6132)

13. Other Pre Specified Outcome: Hospital Anxiety and Depression Scale (HADS): Depression Total Score Including Outliers
Description: as for outcome 12
Time Frame: Baseline (Day 8, Day 37), Post-dose (Period 1/Day 22, Period 2/Day 51)
Population: FAS. Baseline and Post-dose data for Period 1 and Period 2 summarized as LS Mean.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 22 | 22
scores on a scale | 3.1750 (0.4147) | 3.8705 (0.4147)

14. Other Pre Specified Outcome: Pain Catastrophizing Scale (PCS) Including Outliers
Description: PCS is a participant rated 13-item instrument to measure the presence and severity of catastrophizing. Scored 0 (not at all) to 4 (all the time) to statements such as "When I'm in pain…I worry all the time about whether the pain will end". All 13 statements start with "When I'm in pain…". Total score ranged from 0 to 52; higher scores reflected greater impairment. Baseline and Post-dose data for Period 1 and Period 2 summarized as LS Mean. Any observation with a studentized residual >3 or <-3 was considered an outlier.
Time Frame: Baseline (Day 8, Day 37), Post-dose (Period 1/Day 22, Period 2/Day 51)
Population: FAS
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 22 | 22
scores on a scale | 11.4050 (1.0192) | 12.0041 (1.0192)

15. Secondary Outcome: Short-Form McGill Pain Questionnaire (SF-MPQ): Overall Score Including Outliers
Description: SF-MPQ was completed to assess pain over the past week and to assess present pain and consists of 15 pain descriptors: sensory dimension of pain experience (sum of items 1 to 11) and affective dimension (sum of items 12 to 15). Each descriptor was ranked by the participant on a 4-point intensity scale (0=none to 3=severe) and totaled in each subclass (sensory range 0 to 33; affective range 0 to 12). Total (overall) score was sum of items 1 to 15, range 0 to 45; higher scores indicated higher pain/impact. Any observation with a studentized residual >3 or <-3 was considered an outlier.
Time Frame: Baseline (Day 8, Day 37), Post-dose (Period 1/Day 22, Period 2/Day 51)
Population: FAS. Baseline and Post-dose data for Period 1 and Period 2 summarized as LS Mean.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 22 | 22
scores on a scale | 10.0862 (1.2657) | 11.2774 (1.2657)

16. Secondary Outcome: Sphygmomanometry Evoked Allodynia in Relation to the Blood Pressure (BP) Value at Which Allodynia Was Evoked
Description: BP cuff evoked allodynia assessed based on participant response to the following question "When I take your blood pressure, tell me if the cuff's pressure is painful". A standard BP cuff was inflated at approximately 10 millimeters of mercury (mm Hg) per second up to 180 mm Hg or to point when participant experienced pain; performed 3 times on each arm whether or not pain was reported. If no pain elicited at 180 mm Hg, it was recorded that no sphygmomanometry-evoked allodynia occurred. If pain was reported, value (in mm Hg) at which pain first occured was recorded for each of the assessments.
Time Frame: Day 58
Population: FAS; N=number of participants with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- All Study Treatment: Pregabalin, Placebo: Pregabalin administered in Period 1 (75 mg BID Period 1/Day 9 to 11; then 150 mg BID Period 1/Day 12 to 16; then 200 mg BID Period 1/Day 17 to 19; then 225 mg BID Period 1/Day 20 to 22) or administered in Period 2 (75 mg BID Period 2/Day 38 to 40; then 150 mg BID Period 2/Day 41 to 45; then 200 mg BID Period 2/Day 46 to 48; then 225 mg BID Period 2/Day 49 to 51); then taper Period 2/Day 52 to 58.
  Placebo to match study treatment administered in Period 1 or Placebo to match study treatment administered in Period 2.
Arm/Group | All Study Treatment: Pregabalin, Placebo
Number analyzed (Participants) | 12
mm Hg
  Mean Left Arm BP Cuff Pressure | 107.92 (19.837)
  Mean Right Arm BP Cuff Pressure | 129.31 (19.917)

17. Secondary Outcome: Pain at the Bilateral Epicondyle Tender Points Assessed Using American College of Rheumatology (ACR) Classification Criteria
Description: Participant rated severity of pain upon application of 4 kilograms (kg) pressure via dolorimeter at the bilateral epicondyle tender points (2 tender points, 2 centimeters distal to the epicondyles) described in the American College of Rheumatology (ACR) classification criteria and scored on a 0 (no pain) to 10 (worst possible pain) rating scale. Each arm was to be assessed for any pain (one point on each arm) with the application of pressure.
Time Frame: Day 58
Population: FAS; N=number of participants with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | All Study Treatment: Pregabalin, Placebo
Number analyzed (Participants) | 16
scores on a scale
  Pain Severity Left Epicondyle | 6.25 (2.840)
  Pain Severity Right Epicondyle | 5.72 (2.671)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (all causalities) were reported from the time of first dose of study treatment up to 28 days after last dose of study treatment.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 1/24 | 1/25
Other Adverse Events (participants affected / at risk) | 18/24 | 13/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=24) | Placebo (N=25)
Device material issue (General disorders) | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=24) | Placebo (N=25)
Ear pain (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1
Chest discomfort (General disorders) | 0 | 1
Facial pain (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1
Feeling jittery (General disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Pain (General disorders) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood calcium increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Metabolism and nutrition disorders) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 10 | 2
Headache (Nervous system disorders) | 1 | 2
Somnolence (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Euphoric mood (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.